CLINICAL TRIAL: NCT05175547
Title: Clevidipine Infusion for Blood Pressure Management After Successful Revascularization in Acute Ischemic Stroke (CLEVER)
Brief Title: Clevidipine Infusion for Blood Pressure Management After Successful Revascularization in Acute Ischemic Stroke
Acronym: CLEVER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ProMedica Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLEVER
Record Dates: First submitted 2021-11-23; First posted 2022-01-03 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Stroke, Acute; Blood Pressure; Mechanical Thrombectomy
MeSH Terms: conditions — Stroke | interventions — clevidipine

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomized 1:1 to a systolic blood pressure goal after successful MT (mTICI 2c or greater) of either: 90-120 or 90-160mmHg.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intensive blood pressure management group (Active Comparator): Target blood pressure of 90-120mmHg (Intensive BP management group)
  Interventions: Drug: Clevidipine
- Standard blood pressure management group (Active Comparator): Target blood pressure of 90-160mmHg (Standard BP management group)
  Interventions: Drug: Clevidipine

INTERVENTIONS:
Drug: Clevidipine — Blood pressure management with Clevidipine

SUMMARY:
The CLEVER Study is a prospective, 2-arm, randomized, single-center pilot study to assess the safety and efficacy of intensive blood pressure control using Clevidipine (on-label use) in AIS patients undergoing standard of care mechanical thrombectomy (MT) within 24-hours of symptoms onset.

DETAILED DESCRIPTION:
The CLEVER Study is a prospective, 2-arm, randomized, single-center pilot study to assess the safety and efficacy of intensive blood pressure control using Clevidipine (on-label use) in AIS patients undergoing standard of care mechanical thrombectomy (MT) within 24-hours of symptoms onset. Eligible patients will be randomized 1:1 to a systolic blood pressure goal after successful MT (mTICI 2c or greater) of either: 90-120mmHg (Intensive BP management group) or 90-160mmHg (Standard BP management group). Patients enrolled into the study will be followed and assessed for up to 3 months.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18 or older
* 2. Acute hypertension (systolic blood pressure of greater than 140 mmHg) at recanalization
* 3. Anterior circulation ischemic stroke symptoms and confirmed occlusion (ICA, M1, or M2) on angiogram with mechanical thrombectomy initiated within 24 hours since last known well
* 4. Success revascularization score of mTICI 2c or higher after mechanical thrombectomy
* 5. ASPECTS score of greater than 6
* 6. Premorbid mRS 0-4
* 7. Signed informed consent within 30 minutes from end of MT procedure.

Exclusion Criteria:

* 1. Presence of any hemorrhage and/or ASPECT score ≤6 on baseline head CT scan
* 2. Pregnant or lactating
* 3. Acute traumatic brain injury
* 4. Patient on active dialysis
* 5. Intracranial neoplasm
* 6. Acute or recent STEMI in the last 30 days
* 7. Severe arrhythmias, unstable cardiac function
* 8. Any terminal medical condition with life expectancy less than 6 months
* 9. Concurrent enrollment in another trial that could confound the results of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-10-30 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint (Drug-related) | Time from drug initiation to target blood pressure, up to 24 hours after study drug adminstration
  Time to target blood pressure
Primary Safety Endpoint (Disease-related) | 24 hours from the time of treatment with Clevidipine
  Incidence of any hemorrhagic conversion at 24 hours

SECONDARY OUTCOMES:
Drug-related | Up to 24 hours after study drug adminstration
  The efficacy of Clevidipine in maintaining BP within range using area under the curve (AUC) analysis of BP excursions beyond predetermined upper and lower limits using statistical models from the ECLIPSE Trials.
Drug-related, Rate of hypotension requiring intervention | Up to 24 hours after study drug adminstration
  Rate of hypotension requiring intervention
Drug-related, Rate of hypotension and severe hypertension | Up to 24 hours after study drug adminstration
  Rate of hypotension and severe hypertension
Disease-related, Incidence of symptomatic intracerebral hemorrhage | Within 24 hours of randomization
  Incidence of symptomatic intracerebral hemorrhage (sICH), defined as any intracranial hemorrhage and neurologic worsening of at least 4 points on the National Institute of Health Stroke Scale (NIHSS), according to the 2nd European-Australasian Acute Stroke Study (ECASS II) criteria within 24 hours of randomization
Disease-related, Delayed ICH after 24 hours | Within 24 hours of randomization
  Delayed ICH after 24 hours
Disease-related, Incidence of acute kidney injury | From drug adminstration to 90 days post-randomization
  Incidence of acute kidney injury
Disease-related, | 90 days after randomization
  Mortality rate at 90 days
Disease-related, Length of hospital stay | Day 6 (+/- 1 day) post-randomization or discharge (whichever sooner)
  Length of hospital stay
Disease-related, Use of additional hypertensive agents | Up to 24 hours after study drug adminstration
  Use of additional hypertensive agents
Disease-related, Onset of atrial fibrillation or cardiovascular events | Up to 24 hours after study drug adminstration
  Onset of atrial fibrillation or cardiovascular events
Disease-related, mRS 0-2 or return to baseline at 90 days | 90 days post-randomization
  mRS 0-2 or return to baseline at 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Mouhammad Jumaa, MD, Principal Investigator — ProMedica Health System
Locations (1):
- ProMedica Toledo Hospital, Toledo, Ohio, United States

IPD SHARING:
Plan to Share IPD: No